CLINICAL TRIAL: NCT03629366
Title: Supported Employment for Refugees
Acronym: SER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 811270
Record Dates: First submitted 2018-07-09; First posted 2018-08-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Refugees
Keywords: Refugees; Supported Employment; Individual Placement and Support; Employment; Vocational Rehabilitation; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Employment, Supported; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supported Employment (SE) (Experimental): Follow-up with Supported Employment (SE), provided by a job specialist trained in the eight evidence-based principles of Individual Placement and Support (IPS). The SE intervention is provided in addition to the mandatory introduction program for refugees in Norway (treatment as usual).
  Interventions: Behavioral: Supported Employment (SE)
- Treatment as usual (TAU) (Active Comparator): Follow-up with treatment as usual, which involves participation in the mandatory introduction program provided for all refugees in Norway. The program includes training in Norwegian language and culture, as well as the various traditional employment schemes offered by the Norwegian labor and welfare Administration.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Supported Employment (SE) — Supported Employment
  Arms: Supported Employment (SE)
Behavioral: Treatment as usual (TAU) — Treatment as usual
  Arms: Treatment as usual (TAU)

SUMMARY:
Humanitarian crises related to the Syrian conflict have led to a large increase in refugees in Europe in the recent years. There is need for effective approaches to increase labor market participation among refugees, and to reduce the impact of unfavorable exclusion mechanisms among this group. The Supported Employment for Refugees (the SER-trial) is a randomized controlled trial investigating the effectiveness of Supported Employment (SE) for newly arrived refugees who are involved in the mandatory introduction program provided for all refugees in Norway. SE is an intervention that has proved effective in promoting competitive employment among patients with severe mental illness in over twenty international randomized controlled trials, and is currently being evaluated for various new patient groups in ongoing trials. The SER-trial is however the first trial to evaluate the effect of SE for the target group of refugees (who may or may not have mental illness).

ELIGIBILITY:
Inclusion Criteria:

* Refugees in the city of Bergen, Norway
* Expressed desire to work
* Able to have a simple conversation in Norwegian or English

Exclusion Criteria:

* No expressed desire to work
* Unable to have a simple conversation in Norwegian or English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Competitive employment (register data and log books) | 12 months
  Competitive employment will be assessed using register data from the State Register of Employers and Employees. Analyses will be carried out using both intention-to-treat and per protocol analyses. For per protocol analyses, log books from the service providers in the intervention group will be used.

SECONDARY OUTCOMES:
Acculturation (survey data) | 12 months
  Acculturation will be assessed using the Vancouver Index of Acculturation (VIA)
Psychological distress (survey data) | 12 months
  Psychological distress will be assessed using the Hopkins Symptom Checklist-25 (HSCL-25)
Posttraumatic stress (survey data) | 12 months
  Posttraumatic stress will be assessed using the PTSD Checklist for DSM-5 (PCL-5)
Global well-being (survey data) | 12 months
  Global well-being will be assessed using a 10-point Cantril Ladder Scale
Health-related quality of life (survey data) | 12 months
  Health-related quality of life will be assessed using the Euro-Qol Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Vigdis Sveinsdottir, PhD, Principal Investigator — NORCE Norwegian Research Centre; Tonje Fyhn, Principal Investigator — NORCE Norwegian Research Centre
Locations (1):
- NORCE Norwegian Research Centre, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No